CLINICAL TRIAL: NCT03189784
Title: Mobilization With Movement Treatment in Patients With Chronic Ankle Instability
Brief Title: Ankle Instability Treatment in Patients With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, DAVID CRUZ DÍAZ, Physiotherapy coordinator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ankle ujaen
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobilization group (Experimental): this group will receive mobilization with movement techniques.
  Interventions: Other: mobilization with movement techniques
- Control group (No Intervention): The control group will receive no intervention

INTERVENTIONS:
Other: mobilization with movement techniques — patient will receive an anteroposterior stimuli in the talus in order to restore the range of motion
  Other Names: Joint mobilizations
  Arms: mobilization group

SUMMARY:
Ankle joint self mobilization.

DETAILED DESCRIPTION:
The intervention would consist in the administration of self mobilization with movement techniques in patients with chronic ankle instability in addition to an exercise program

ELIGIBILITY:
Inclusion Criteria:

* ankle range of motion limitation respect the contralateral ankle.
* At least two episodes of giving way on the affected ankle.
* Scores of at least 24 in the cumberland ankle instability tool.

Exclusion Criteria:

* recent fractures of the involved limb.
* Vestibular or balance dysfunction.
* Acute ankle sprain.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
range of motion | from baseline prior to the beginning of the intervention to the completion of the study at four weeks.
  the ankle range of motion will be measured by goniometry.

SECONDARY OUTCOMES:
dynamic balance | from baseline prior to the beginning of the intervention to the completion of the study at four weeks.
  Dynamic balance will be determined by the star excursion balance test
Self reported instability | from baseline prior to the beginning of the intervention to the completion of the study at four weeks.
  Self reported instability will be assessed by the Cumberland ankle instability tool

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - University of Jaen campus, Jaén
  - University of Jaen, Jaén

IPD SHARING:
Plan to Share IPD: No